CLINICAL TRIAL: NCT06624189
Title: Active Choice Clinical Decision Support: Hepatocellular Carcinoma Screening in Patients With Cirrhosis
Brief Title: Active Choice Clinical Decision Support (CDS): Hepatocellular Carcinoma (HCC) Screening in Patients With Cirrhosis
Status: Enrolling by invitation | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: QI-Active Choice CDS
Record Dates: First submitted 2024-10-01; First posted 2024-10-02 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Hepatocellular Carcinoma; Cirrhosis
MeSH Terms: conditions — Carcinoma, Hepatocellular; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention: Auto-pended bot liver ultrasound order: Participants in the intervention group will receive an auto-pended bot liver ultrasound order that will prompt providers at the time of encounter to place appropriate imaging orders for hepatocellular carcinoma (HCC) screening.
  Interventions: Other: Auto-pended bot liver ultrasound order
- Control: Usual Care: Participants in the control group will not receive the auto-pended bot liver ultrasound order.

INTERVENTIONS:
Other: Auto-pended bot liver ultrasound order — This alert prompt providers at the time of encounter to place appropriate imaging orders for hepatocellular carcinoma (HCC) screening in patients with cirrhosis.
  Groups: Intervention: Auto-pended bot liver ultrasound order

SUMMARY:
The research team will evaluate the effectiveness of an auto-pended bot liver ultrasound order that will prompt providers at the time of encounter to place appropriate imaging orders for hepatocellular carcinoma (HCC) screening in patients with cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* cirrhosis diagnosis,
* 6 months or more after since most recent imaging.

Exclusion Criteria:

* previous liver transplant,
* HCC diagnosis,
* receiving hospice care,
* completed external imaging in the past 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with a cirrhosis diagnosis, and at the date of their appointment had been 6 months or more after their most recent imaging.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2026-04-24 (Estimated); Study Completion 2026-07-24 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants for whom the Physician Completed Ordering of the Pending Liver Ultrasound | Day 1

SECONDARY OUTCOMES:
Percentage of Participants with Completed Liver Ultrasound Imaging | Day 1
HCC Diagnosis Rate from Completed Liver Ultrasound Imaging | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Saul Blecker, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
This is a quality improvement (QI) project and individual participant data (IPD) will not be shared with other researchers.